CLINICAL TRIAL: NCT03813732
Title: the Effect of Using the Tyransconjunctival Approach Alone Versus Using Transconjunctival Approach Together With Lateral Canthotomy in Orbital Fractures
Brief Title: Using the Transconjuctival Approach Alone Versus Using it Together With Lateral Canthotomy in Orbital Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nashwa Osama, assistant researcher in national research centre, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-01-03
Record Dates: First submitted 2019-01-09; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Orbital Fractures
Keywords: trans-conjunctival approach
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Intervention Model Description: 1. Pre-operative phase:
     Patients will be subjected to:
     1. Case history including personal data, medical, surgical and family history.
     2. Clinical examination.
     3. Preoperative anesthesia assessment for fitness for general anesthesia.
     4. Treatment planning.
  2. Operative phase:
     All cases will undergo surgery under general anesthesia.
  3. Postoperative care:
     Proper postoperative instructions will be given the patient, in addition to the postoperative medications including antibiotics, corticosteroids and analgesics.
  4. Postoperative evaluation and follow-up:
  12) Outcomes: outcome Method of measurement Measuring unit Primary outcome Assessment of the esthetics. Visual analog scale Numerical Secondary outcome pain Visual analog scale Numerical (1-10)
Masking Description: Outcomes:
  outcome Method of measurement Measuring unit Primary outcome Assessment of the esthetics. Visual analog scale Numerical Secondary outcome pain Visual analog scale Numerical (1-10)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orbital fracture (Other): using the trans-conjunctival approach with lateral canthotomy
  Interventions: Procedure: orbital fracture

INTERVENTIONS:
Procedure: orbital fracture — using the trans-conjunctival approach alone in restoring the esthetics compared with using it along in addition to lateral canthotomy which is important in providing wider surgical area

SUMMARY:
All cases will undergo surgery under general anesthesia. Evaluation of patients with suspected orbital fracture should involve radiologic examination, motility test, diplopia field test and exophthalmometry. Plain X-ray films, although rarely used, with the Caldwell and Waters view may be done as a screening evaluation for possible fractures and foreign bodies. An orbital computed tomography, the gold standard in trauma, CT with contiguous thin axial and coronal sections should be ordered to confirm the diagnosis and plan for treatment

Postoperative care:

Proper postoperative instructions will be given the patient, in addition to the postoperative medications including antibiotics, corticosteroids and analgesics.

DETAILED DESCRIPTION:
This study will be carried out on patients attending the outpatient clinic in Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Cairo University.

10. Eligibility criteria:

* Inclusion criteria:
* Age group: from 15 to 60 years old.
* Patients with pure blow-out fractures.
* Exclusion criteria:

  * Patients suffering from dermatological diseases,

    11. Interventions:
    1. Pre-operative phase:

       Patients will be subjected to:
       1. Case history including personal data, medical, surgical and family history.
       2. Clinical examination.
       3. Preoperative anesthesia assessment for fitness for general anesthesia.
       4. Treatment planning.
    2. Operative phase:

       All cases will undergo surgery under general anesthesia. The inferior wall can be easily accessed through transcutaneous or transconjunctival approach (with or without lateral canthotomy). The latter avoids a visible scar and is less likely to result in eyelid retraction. The medial wall can be accessed through transcaruncular approach. Careful exploration under the periosteum allows easy visualization of the fracture boundaries as well as correction of the herniated tissue.

       Then various implants can be used to support the orbital soft tissue and prevent recurrent herniation. Porous polyethylene sheets (Medpor) are one of most commonly used implant materials. Other autogenous (cranial, rib or iliac bone graft) or alloplastic (gelatin film, silicone sheet, Teflon, Supramid, titanium mesh or bioresorbable copolymer plates) materials are also available.

       Periocular fractures are often managed first by the ophthalmologist. With good clinical examination and radiographic imaging, an informed decision can be made whether surgical intervention is required.
    3. Postoperative care:

Proper postoperative instructions will be given the patient, in addition to the postoperative medications including antibiotics, corticosteroids and analgesics.

ELIGIBILITY:
* Inclusion criteria:
* Age group: from 15 to 60 years old.
* Patients with blow-out fractures.
* Exclusion criteria:

  * Patients suffering from dermatological diseases,

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of the esthetics | 3 months
  Visual analog scale numerical1-10

SECONDARY OUTCOMES:
Infection | 3month
  Accent/present

CONTACTS AND LOCATIONS:
Locations (1):
- Alasr elany, Giza, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee HB, Lee SH. New anthropometric data for preoperative planning in orbital wall fracture treatment: the use of eyelid drooping. Arch Craniofac Surg. 2018 Dec;19(4):248-253. doi: 10.7181/acfs.2018.02096. Epub 2018 Dec 27. PMID 30613085